CLINICAL TRIAL: NCT06505070
Title: The Effect of Recreational Games on Happiness, Life Satisfaction, Loneliness, and Somatisation in Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Duzce-U-merve0003
Record Dates: First submitted 2024-07-02; First posted 2024-07-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Happiness; Life Satisfaction; Loneliness; Somatization
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Individuals in the control group continued their daily routines. They were chosen from another nursing home to avoid interaction with the experimental group.
- Experimental group (Experimental): Participants in the intervention group engaged in bingo, matching pairs, word challenges, and hot-and-cold games, organized into groups of eight individuals. They adhered to the game instructions and participated in sessions twice a week for 2 months, totalling 16 sessions. In each session, all individuals played all four games, so one played 64 games in 16 sessions. Sessions are planned to last 45 minutes.
  Interventions: Behavioral: Recreational Games

INTERVENTIONS:
Behavioral: Recreational Games — 40 individuals in the intervention group were introduced to 15 games. Researchers conducted these sessions and provided participants with instructions and rules for the games. Then, they were asked to rate the games from 1 to 10. In this form, the elderly individuals evaluated the games by determining the minimum "1" and maximum "10" points according to their interest and willingness to play. Thus, it was ensured that individuals freely choose the games they want to play. As a result, bingo, matching pairs, word challenges and hot-cold games, which received the highest scores from the participants, were selected to be played.
  Arms: Experimental group

SUMMARY:
As per the United Nations population projections, the percentage of individuals aged 65 and older in the global population is expected to increase from 10% in 2022 to 16% by the year 2050. In response to this demographic shift, the United Nations emphasizes the importance of ageing countries establishing long-term sustainable care institutions and taking measures to ensure the adaptation of the elderly to these institutions. Recreational activities play a crucial role in supporting and encouraging elderly individuals to maintain active and productive lives in their old age while preserving their social roles.

Aim: To measure the influence of recreational games on somatisation, loneliness, happiness and life satisfaction among elderly individuals.

DETAILED DESCRIPTION:
As per the United Nations population projections, the percentage of individuals aged 65 and older in the global population is expected to increase from 10% in 2022 to 16% by the year 2050. In response to this demographic shift, the United Nations emphasizes the importance of ageing countries establishing long-term sustainable care institutions and taking measures to ensure the adaptation of the elderly to these institutions. Recreational activities play a crucial role in supporting and encouraging elderly individuals to maintain active and productive lives in their old age while preserving their social roles.

Aim: To measure the influence of recreational games on somatisation, loneliness, happiness and life satisfaction among elderly individuals.

Method: This study employed a nonrandomized experimental design featuring pretest-posttest control groups. The study was conducted across two distinct nursing homes to prevent potential influence between individuals in the control and intervention groups.

The research was conducted from April to August 2018 within two nursing homes in Turkey. Inclusion criteria comprised individuals meeting the following conditions: 1) aged 65 years and above and residing in the designated nursing homes during the study duration; 2) expressing willingness to participate in the research; 3) attaining a score of 23 or higher (for individuals with five or more years of formal education) or 19 or higher (for those with fewer than five years of formal education) on the Standardized Mini-Mental State Examination for Educated and Uneducated Individuals (SMMSE); and 4) displaying openness to communication.

A power analysis, executed utilizing the G Power 3.0.10 software, determined the requisite number of participants for both the intervention and control groups. Given a type I error rate of 0.05, a type II error rate of 0.80, and an effect size of 0.5, it was established that a minimum of 27 participants were needed for each group. Considering the potential occurrence of missing data during the study, 40 participants meeting the inclusion criteria were applied to participants in both groups.

Data collection tools: The Standardized Mini-Mental State Examination for Educated and Uneducated Individuals (SMMSE) was utilized to ascertain the eligibility of older individuals for participation in the study. Data were collected utilizing a Personal Information Form, the Oxford Happiness Questionnaire Short Form (OHQ-S), the Satisfaction with Life Scale (SWLS), the De Jong Gierveld Loneliness Scale (DJGLS), and the Symptom Check-List Somatisation Subscale (SCL-90-R).

Game selection: After an extensive literature review, the researcher identified 15 games. These games were introduced to participants in the intervention group, enabling them to make informed selections subsequent to receiving instructions.

Interventions: Residents of the nursing homes where the study took place were informed about the research. The SMMSE was administered to individuals who expressed interest in taking part.

Application of pre-tests: OHQ-S, DJGLS, SWLS, and SCL-90-R were applied to a total of 80 individuals in both nursing homes who met the study inclusion criteria.

Selection of the games to be included in the application: One nursing home was allocated as the intervention group to minimize potential interaction between the groups, while the other was designated as the control group. During two sessions, 40 individuals in the intervention group were introduced to 15 games. Researchers conducted these sessions and provided participants with instructions and rules for the games. Then, they were asked to rate the games from 1 to 10. In this form, the elderly individuals evaluated the games by determining the minimum "1" and maximum "10" points according to their interest and willingness to play. Thus, it was ensured that individuals freely choose the games they want to play. As a result, bingo, matching pairs, word challenge and hot-cold games, which received the highest scores from the participants, were selected to be played.

Preparing the playground and organizing the groups: For the elderly to play games, a room on the ground floor of the institution with a sun-drenched, spacious sliding door opening to the garden was preferred. Five groups of 8 people were formed for the games. These groups were determined according to their wishes, taking into account the available hours of the elderly individuals. When one group completed the games, 15-20 minute breaks were given for that group to leave the room and for the other group to gather and prepare for the games.

Playing games: Participants in the intervention group engaged in bingo, matching pairs, word challenges, and hot-and-cold games, organized into groups of eight individuals. They adhered to the game instructions and participated in sessions twice a week for 2 months, totalling 16 sessions. The groups were formed by the requests of the participants, considering their available time. In each session, all individuals in the group played all four games, so one individual played 64 games in a total of 16 sessions. Sessions are planned to last 45 minutes.

Application of posttests: Individuals in the groups underwent administration of OHQ-S, DJGLS, SWLS, and SCL-90-R at two consecutive intervals: 1 week (post-test) and 1 month (follow-up-test) after the conclusion of the game.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years and above and residing in the designated nursing homes during the study duration,
* expressing willingness to participate in the research,
* attaining a score of 23 or higher (for individuals with five or more years of formal education) or 19 or higher (for those with fewer than five years of formal education) on the Standardized Mini-Mental State Examination for Educated and Uneducated Individuals,
* displaying openness to communication.

Exclusion Criteria:

* Unconscious
* Individuals who decline to participate in the study
* Individuals using antipsychotic medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Happiness levels | Before the interventions (pre-test), 1 week (post-test) and 1 month (follow-up test) after the interventions
  Oxford Happiness Questionnaire Short Form: The form, created by Hills and Argyle, comprises a 29-item scale utilizing a 6-point Likert-type scoring system. Its abbreviated version, containing 7 items, was translated into Turkish in 2011. The internal consistency, evaluated using Cronbach's alpha, resulted in a value of 0.74, whereas the test-retest reliability coefficient was recorded as 0.85. The highest score that can be obtained from the scale is 174 and the lowest score is 29. An increase in the score means an increase in the level of happiness.
Satisfaction with life levels | Before the interventions (pre-test), 1 week (post-test) and 1 month (follow-up test) after the interventions
  Satisfaction with Life Scale: The scale was developed by Diener et al. (1985) to determine the satisfaction people get from life and consists of a 7-point Likert scale with unidimensional structure comprising 5 items. During its adaptation to the Turkish language, the scale underwent modification into a 5-point Likert scale. The Cronbach alpha of the scale was 0.88 and the test-retest reliability coefficient was 0.97.
Loneliness levels | Before the interventions (pre-test), 1 week (post-test) and 1 month (follow-up test) after the interventions
  De Jong Gierveld Loneliness Scale: The scale, crafted by Gierveld and Kamphuis (1985) to gauge the degree of loneliness among older individuals, underwent linguistic adaptation to Turkish in 2015. The scale's Cronbach alpha was 0.85. Comprising 11 items and 2 subscales, the scale encompasses six negative items evaluating emotional loneliness and 5 positive items appraising social loneliness. Employing a 3-point Likert-type scale, with five items scored inversely, the scale's minimum and maximum scores are 0 and 22, respectively.
Somatisation levels | Before the interventions (pre-test), 1 week (post-test) and 1 month (follow-up test) after the interventions
  Symptom Check-List Somatisation Subscale: The scale, originally developed by Derogatis, Lipman, and Covi (1973) and subsequently adapted to the Turkish language by Kılıc (1991), is known as SCL-90-R. It is a diagnostic tool for assessing psychological concerns and identifying individual symptoms. The scale comprises nine subcategories, which encompass interpersonal sensitivity, obsessive-compulsive behaviour, somatisation, paranoid ideation, psychoticism, anger-hostility, anxiety, depression and phobic anxiety, utilizing a 4-point Likert type scale. The reliability coefficient for the somatisation subcategory was found to be 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Hasibe Kadıoglu, Study Director — Marmara University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

REFERENCES:
- [Derived] Cakar M, Kadioglu H. The effect of recreational games on happiness, life satisfaction, loneliness, and somatisation in elderly individuals: a non-randomized controlled trial. BMC Psychol. 2025 Mar 22;13(1):289. doi: 10.1186/s40359-025-02583-6. PMID 40121499